CLINICAL TRIAL: NCT07323420
Title: A Clinical Study on the Effects of Different Inspiratory:Expiratory Ratios on Respiratory Function and Recovery in Pediatric Patients Undergoing Dental Procedures Under General Anesthesia
Brief Title: Effects of Different Inspiratory:Expiratory Ratios on Respiratory and Recovery Outcomes During Dental Procedures Under General Anesthesia in Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Gözde Nur Erkan, Assistant Professor, Kırıkkale University
Other Study IDs: KU-ERKAN-004
Record Dates: First submitted 2025-11-14; First posted 2026-01-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Function; Pediatric Anesthesia; General Anesthesia
Keywords: General Anesthesia; Anesthesia Recovery; Emergence from Anesthesia; Mechanical Ventilation; I:E Ratio; Recovery Quality
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Control: Patients who emerge from anesthesia earlier than planned without pre-emergence preparation. A minimum of 15 patients will be enrolled in this group.
- Group 2: I:E 1:2: Patients undergoing standart dental procedures under general anesthesia; during the last phase of the procedure, mechanical ventilation will be applied with an I:E ratio of 1:2. A minimum of 30 patients will be enrolled in this group.
- Group 3: I:E 1:3: Patients undergoing standart dental procedures under general anesthesia; during the last phase of the procedure, mechanical ventilation will be applied with an I:E ratio of 1:3. A minimum of 30 patients will be enrolled in this group.

SUMMARY:
This observational study aims to evaluate the effects of different inspiratory to expiratory (I:E) ratios (1:2 vs. 1:3) during mechanical ventilation in pediatric patients undergoing dental procedures under general anesthesia. Due to behavioral challenges, dental phobia, or medical conditions, general anesthesia is often required to ensure immobility and cooperation during dental treatments in children.

In the clinic where the study will be conducted, the I:E ratio is routinely adjusted approximately 20-30 minutes before the end of the procedure to facilitate a smoother transition to spontaneous breathing during emergence from anesthesia. While 1:2 is commonly used, the 1:3 ratio may improve respiratory efficiency and recovery by prolonging the expiratory phase.

The study aims to compare vital signs, respiratory parameters (heart rate, blood pressure, SpO₂, EtCO₂, respiratory rate), recovery quality, and respiratory complications between the two I:E ratios. The findings aim to optimize ventilation strategies and improve patient comfort and safety during emergence from anesthesia.

DETAILED DESCRIPTION:
The recent study involves pediatric patients undergoing dental procedures under general anesthesia following routine and standard clinical protocols. No additional interventions beyond standard care will be applied.

Specifically for the study, a non-invasive, observational scoring system will be used during the emergence phase to assess respiratory quality without requiring any extra tests or procedures. The scoring includes observation of spontaneous breathing, accessory muscle use, airway patency, physical responses to painful stimuli, and coughing episodes.

Patients will receive the same anesthesia and dental treatment as those not included in the study. The study compares the effects of routine inspiratory:expiratory (I:E) ratios used during mechanical ventilation on respiratory and recovery outcomes.

Variables assessed include vital and respiratory parameters (heart rate, blood pressure, SpO₂, EtCO₂, respiratory rate, peak airway pressure, time to spontaneous breathing, and physical/hemodynamic responses during spontaneous breathing), respiratory quality post-extubation (evaluated via the study-specific scale), and recovery parameters (physical responses during airway suctioning/extubation, presence of bronchospasm/ laryngospasm, agitation levels measured preoperatively by Modified Yale Preoperative Anxiety Scale and postoperatively by the Pediatric Anesthesia Emergence Delirium Scale (PAED), Modified Aldrete score, and discharge times from recovery and hospital wards).

All data will be recorded in a patient tracking form prepared for the study. Induction, maintenance, emergence from anesthesia, and management of any complications will follow routine clinical practice without any changes. No modifications to anesthesia or dental treatment protocols will be required for the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients scheduled for dental procedures under general anesthesia at our faculty.
* American Society of Anesthesiologists (ASA) Physical Status I or II.
* Age between 2 and 12 years.
* Written informed consent obtained from parents or legal guardians.

Exclusion Criteria:

* Patients whose parents or legal guardians decline participation.
* Presence of adenoid hypertrophy >30%.
* Macroglossia or retrognathia.
* Severe obesity or developmental delay.
* History of delayed emergence from anesthesia.
* ASA Physical Status III or higher.
* Anesthesia duration less than 1 hour or more than 3 hours.
* Patients with difficult airway management or ventilation.
* Known pulmonary or airway diseases or anomalies.
* Use of pharmacological agents that may affect spontaneous respiratory quality.
* Presence of neuromuscular disorders affecting respiratory function.
* Age <2 years or >12 years.
* Administration of medications intraoperatively or preoperatively that may influence respiratory dynamics during emergence (e.g., atropine, lidocaine, steroids).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include pediatric patients aged 2 to 12 years who are scheduled to undergo routine dental procedures under general anesthesia at our faculty. Eligible participants are classified as American Society of Anesthesiologists (ASA) Physical Status I or II. Patients with airway anomalies, significant adenoid hypertrophy, macroglossia, retrognathia, severe obesity, developmental delays, or a history of delayed emergence from anesthesia will be excluded. Children requiring anesthesia for less than 1 hour or more than 3 hours, those with known pulmonary or airway diseases, neuromuscular disorders affecting respiration, or receiving medications that could alter spontaneous breathing during emergence (e.g., atropine, lidocaine, steroids) are also excluded. Written informed consent must be obtained from parents or legal guardians prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Post-Extubation Respiratory Quality | During 10 minutes after extubation
  Respiratory quality will be assessed using a study-specific observational scale (range 0-10; higher scores indicate poorer respiratory quality). Components include spontaneous breathing adequacy, accessory muscle use, airway patency, response to painful stimuli, and coughing episodes.
Respiratory Rate (RR) | During the emergence preparation period (approximately 25-35 minutes prior to extubation, up to 40 minutes if required)
  Mean respiratory rate (breaths/min) recorded during spontaneous breathing while EtCO₂ is maintained within the standardized target range, for each I:E ratio group (1:2 vs. 1:3).
Peak Airway Pressure (PeakP) | During the emergence preparation period (approximately 25-35 minutes prior to extubation, up to 40 minutes if required)
  Peak airway pressure (cmH₂O) recorded during emergence preparation period for each I:E ratio group (1:2 vs. 1:3).
Heart Rate | During the emergence preparation period (approximately 20-30 minutes prior to extubation, up to 40 minutes if required)
  Mean heart rate (beats/min) recorded during spontaneous breathing while EtCO₂ and sevoflurane MAC are maintained within the standardized target range, for each I:E ratio group (1:2 vs. 1:3).
Blood Pressure | During the emergence preparation period (approximately 20-30 minutes prior to extubation, up to 40 minutes if required)
  Mean arterial blood pressure (mmHg) recorded during spontaneous breathing while EtCO₂ and sevoflurane MAC are maintained within the standardized target range, for each I:E ratio group (1:2 vs. 1:3).

SECONDARY OUTCOMES:
Physical Response During Extubation | From 2 minutes before extubation to 2 minutes after extubation
  The patient's physical response during removal of the endotracheal tube will be assessed by direct observation at the time of extubation. Responses will be evaluated once during the extubation process based on the presence of facial grimacing, upper extremity movement, lower extremity movement, or other observable involuntary motor responses.
Occurrence of Bronchospasm or Laryngospasm | From extubation until 30 minutes after extubation
  The occurrence of bronchospasm or laryngospasm during or immediately after extubation will be recorded. These events will be identified based on clinical signs such as increased airway resistance, wheezing, stridor, oxygen desaturation, or the need for medical intervention.
Preoperative Anxiety Level Assessed by the Modified Yale Preoperative Anxiety Scale (mYPAS) | Immediately before surgery (prior to operating room entry)
  Preoperative anxiety will be assessed using the Modified Yale Preoperative Anxiety Scale (mYPAS), which ranges from 23 to 100, with higher scores indicating greater levels of anxiety. The assessment will be performed before anesthesia induction.
Pediatric Anesthesia Emergence Delirium (PAED) Score | From emergence from anesthesia through recovery unit stay until discharge, assessed up to 1 hour
  The Pediatric Anesthesia Emergence Delirium (PAED) scale is a validated observational tool used to assess the presence and severity of emergence delirium in pediatric patients after anesthesia. The scale consists of five items, with total scores ranging from 0 to 20, where higher scores indicate more severe emergence delirium.
Modified Aldrete Score | From emergence from anesthesia through recovery unit stay until discharge, assessed up to 1 hour
  The Modified Aldrete Score assesses postoperative recovery, including activity, respiration, circulation, consciousness, and oxygen saturation. Total scores range from 0 to 10, with higher scores indicating more complete recovery.
Postoperative transfer times | From end of surgery until transfer to the hospital ward, assessed up to 2 hours
  Operating Room → Recovery Room: Time (in minutes) from the end of surgery to patient transfer from the operating room to the recovery room.
  Recovery Room → Hospital Ward: Time (in minutes) from patient arrival in the recovery room to transfer to the hospital ward.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Faculty of Dentistry, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be publicly shared; however, the dataset will be made available upon reasonable request to the corresponding author, subject to approval and relevant ethical considerations.